CLINICAL TRIAL: NCT04812509
Title: A Multi-center, Randomized, Double-blind, Parallel Controlled Phase Ⅲ Clinical Study to Evaluate the Efficacy and Safety of Recombinant Human Anti RANKL Monoclonal Antibody Injection (MW032) and Denosumab (Xgeva®) in Subjects With Bone Metastases From Solid Tumors
Brief Title: Efficacy and Safety of MW032 and Xgeva® in Subjects With Bone Metastases From Solid Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MW032-2019-CP301
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Bone Metastases
Keywords: Denosumab; Biosimilarity; pharmacokinetics; pharmacodynamics; safety
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MW032 (Experimental): MW032 injection(120mg) was administered subcutaneously once every 4 weeks for a maximum of 13 consecutive doses throughout the trial, according to the investigator's assessment.
  Interventions: Drug: MW032
- Xgeva® (Active Comparator): Xgeva® injection(120mg) was administered subcutaneously every 4 weeks for a maximum of 13 cumulative doses throughout the trial,according to the investigator's assessment.
  Interventions: Drug: Xgeva

INTERVENTIONS:
Drug: MW032 — The active ingredient of MW032 is a recombinant human anti-RANKL monoclonal antibody ,subcutaneous injection of 120 mg (1.7ml)every 4 weeks for a maximum of 13 consecutive doses throughout the trial.
  Other Names: recombinant human anti-RANKL monoclonal antibody injection
  Arms: MW032
Drug: Xgeva — The active ingredient of Xgeva® is denosumab,subcutaneous injection of 120 mg (1.7ml)every 4 weeks for a maximum of 13 consecutive doses throughout the trial.
  Other Names: Denosumab Injection
  Arms: Xgeva®

SUMMARY:
A multi-center, randomized, double-blind, parallel controlled Phase III clinical study to evaluate the clinical efficacy and safety of MW032 and Xgeva® in patients with bone metastases from solid tumors.

DETAILED DESCRIPTION:
This is A multi-center, randomized, double-blind, parallel controlled Phase III clinical trial.

The primary objective is to evaluate the clinical efficacy of MW032 and Xgeva® in patients with bone metastases from solid tumors.

The secondary objective are to evaluate the clinical safety and immunogenicity of MW032 and Xgeva® in patients with bone metastases from solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological confirmed malignant tumors (except hematological tumors);
2. Bone metastasis diagnosed by imaging (bone X-ray, CT scanning or magnetic resonance scanning) or pathology (bone biopsy) can be examined within 3 months before signing the informed consent,according to 《The expert consensus on clinical diagnosis and treatment of bone metastases and bone related diseases of malignant tumors (2014)》；
3. No limited of gender,age ≥ 18 years old;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2;
5. Estimated survival time was more than 6 months;
6. Subjects must have adequate organ function at baseline as defined below:① hematology: neutrophils ≥ 1,500/mcL, platelets ≥ 75,000/mcL, hemoglobin ≥ 80 g / L; ② renal function: creatinine (CR) clearance rate ≥ 30 ml / min; ③ Liver function: serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) were less than or equal to 2.0 × upper normal limit (ULN) in subjects without liver metastasis; ALT and AST were less than or equal to 5.0 × ULN in subjects with liver metastasis; serum total bilirubin was less than or equal to 1.5 × ULN; ④ serum calcium (albumin correction) was more than or equal to 2.0 mmol / L (8.0 mg / dl) but less than or equal to 2.9 mmol / L (11.5 mg / dl). Note: calcium supplements should not be used at least 8 hours before serum calcium determination in screening period;
7. Subjects has understood the nature and purpose of the study, as well as the research procedure, and the subject has signed the written informed consent;

Exclusion Criteria:

1. Subjects with diseases not suitable for the study,in the Investigator's opinion (according to the subject's report or medical record review), such as:Other malignant tumors (different from the malignant solid tumors required in this study protocol) occurred within 3 years before enrollment, and in the active period;Other diseases affecting bone metabolism, such as vitamin D deficiency rickets, osteomalacia and primary osteoporosis, hyperparathyroidism, osteitis deformans, etc. (excluding osteoporosis);Human immunodeficiency virus or Treponema pallidum infection;Unstable liver disease, active period of hepatitis B virus or hepatitis C virus infection;Other serious or unstable physical or mental disorders.
2. Brain metastasis.
3. Oral and dental diseases: previous or current evidence of osteomyelitis or necrosis of the jaw; acute dental or mandibular diseases, need to be treated oral surgery; planned invasive dental surgery; failed dental or oral surgery.
4. Subjects with bone metastases need radiotherapy or surgery.
5. Previous treatment with denosumab.
6. Patients who had received any kind of intravenous or oral bisphosphonates before administration of the first study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
uNTx/uCr | from baseline to week 13
  Compare MW032 and Xgeva® for percentage change in bone conversion index (BTM) - urinary type I collagen cross-linked peptide (uNTx) adjusted for urinary creatinine (uCr) in Chinese subjects with solid tumor bone metastasis (uNTx/uCr from baseline to week 13)

SECONDARY OUTCOMES:
uNTx/uCr | from baseline to weeks 5,25,37 and 53
  Compare the percentage change in MW032 and Xgeva® for bone conversion indicator uNTx/uCr among subjects with solid tumor metastasis (from baseline to weeks 5,25,37 and 53).
S-BALP | from baseline to weeks 5,13,25,37 and 53
  Compare the changes of bone specific alkaline phosphatase (S-BALP) from baseline to weeks 5,13, 25,37 and 53.
SRE | from baseline to week 53
  SRE occurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang S, Yin Y, Xiong H, Wang J, Liu H, Lu J, Zhang Q, Zhang L, Zhong J, Nie J, Lei K, Wang H, Yang S, Yao H, Wu H, Yu D, Ji X, Zhang H, Wu F, Xie W, Li W, Yao W, Zhong D, Sun H, Sun T, Guo Z, Wang R, Guo Y, Yu Z, Li D, Jin H, Song H, Chen X, Ma W, Hu Z, Liu D, Guo Y, Tang J, Jiang Z. Efficacy, Safety, and Population Pharmacokinetics of MW032 Compared With Denosumab for Solid Tumor-Related Bone Metastases: A Randomized, Double-Blind, Phase 3 Equivalence Trial. JAMA Oncol. 2024 Apr 1;10(4):448-455. doi: 10.1001/jamaoncol.2023.6520. PMID 38329745